CLINICAL TRIAL: NCT06664775
Title: An Open Label, Prospective, Randomized, Parallel Groups, Multicenter Study to Compare the Efficacy and Safety of TachoSil® Versus Surgicel™ Original (Oxidized Regenerated Cellulose) as an Adjunct to Control Mild to Moderate Soft Tissue Bleeding During Surgery.
Brief Title: A Study to Compare the Efficacy and Safety of TachoSil and Surgicel Original as an Adjunct to Control Mild to Moderate Soft Tissue Bleeding During Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Corza Medical GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CM-TS01
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage | interventions — TachoSil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TachoSil (Experimental)
  Interventions: Biological: TachoSil
- Surgicel Original (Active Comparator)
  Interventions: Biological: Surgicel Original

INTERVENTIONS:
Biological: TachoSil — Adjunct to hemostasis
  Arms: TachoSil
Biological: Surgicel Original — Adjunct to hemostasis
  Arms: Surgicel Original

SUMMARY:
The purpose of this clinical study is to assess the efficacy and safety of TachoSil compared to the widely known and used for > 60 years local hemostatic product Surgicel Original as an adjunct to control mild to moderate soft tissue bleeding during surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Elective open abdominal, retroperitoneal, pelvic, or thoracic surgery. Elective transplant surgery except for liver or heart transplants is included.
2. The participant has a need for secondary hemostatic study intervention at the TBS with mild to moderate bleeding Grade 1 and Grade 2 according to the VIBe Scale.
3. Presence of an appropriate mild to moderate bleeding soft tissue TBS identified intra-operatively by the surgeon.
4. The TBS size < 21 cm2/3.3 in2.
5. Ability to firmly press study intervention at TBS until 3 minutes after randomization.

Exclusion Criteria:

1. Participants undergoing cardiovascular, hepatic, and laparoscopic and robotic surgeries.
2. Congenital or acquired disorders of coagulation.
3. Diseases requiring constant use of any anticoagulant drugs that cannot be safely washed out prior to randomization.
4. Screening Hemoglobin < 9 mg/dL, platelets < 75 × 103/µL, and/or international normalized ratio (INR) > 1.5.
5. Acute major bleeding during surgery.
6. Participant with TBS in an actively infected field.
7. Target bleeding site is from large defects in arteries or veins where the injured vascular wall requires repair with maintenance of vessel patency.
8. Target bleeding site with major arterial bleeding requiring suture or mechanical ligation.
9. Bleeding site is in, around, or in proximity to foramina in bone, or areas of bony confine.
10. Participants with Grade '0', '3', and '4' bleeding at TBS according to VIBe Scale.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Hemostatic success within 3 minutes | within 3 minutes of study intervention
  Proportion of participants achieving hemostatic success at the target bleeding site (TBS) within 3 minutes after application of study intervention

SECONDARY OUTCOMES:
Hemostatic success within 6 minutes | within 6 minutes of study intervention
  Proportion of participants achieving hemostatic success within 6 minutes after application of study intervention
Study intervention failures | within 6 minutes of study intervention
  Proportion of study intervention failures, defined as failure to achieve hemostatic success within 6 minutes after application of study intervention or bleeding requiring additional intervention during the 6 minutes after application of study intervention
hemostatic success from moderate bleeding within 3 minutes | within 3 minutes of study intervention
  Proportion of participants with moderate bleeding achieving hemostatic success at the TBS within 3 minutes after application of study intervention

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Torrance Memorial, Torrance, California
  - St. Anthony Hospital, Lakewood, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - University Of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Washington University, St Louis, Missouri
  - Atrium Health Carolinas Medical Center, Charlotte, North Carolina
  - The Ohio State University Medical Center, Columbus, Ohio